CLINICAL TRIAL: NCT00287144
Title: Observations of Leng Term Effects From Post Partum Thyroiditis.
Brief Title: Post Partum Thyroiditis 2: Long Term Observations
Status: Withdrawn | Type: Observational
Why Stopped: the doctor performing the study suddenly changed work and moved
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Geir Hoff, Head of Dept. of Medicine, Sykehuset Telemark
Other Study IDs: 399702
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples to estimate thyroid function
Oversight: Data Monitoring Committee: No

SUMMARY:
The study tries to determine if post partum thyroiditis has marked long term (20 years after partum) risk for developing hypothyroidism.

DETAILED DESCRIPTION:
This is study where we follow up women who in 1985 were checked for the occurrence of post partum thyroiditis 6 week after labour. The former patients have been invited to participate by answering a questionnaire and by providing results from blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Defined group of women who tested positive for post partum thyroiditis in 1985.
* Control group randomly picked from those who tested negative.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Long-term follow-up of women who developed post-partum thyroiditis within 6 weeks after birth in 1985
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janna Berg, Principal Investigator — Sykehuset Telemark HF, Skien, Norway
Locations (1):
- Sykehuset Telemark HF, Skien, Norway